CLINICAL TRIAL: NCT04042480
Title: A Phase 1 Study of SGN-CD228A in Select Advanced Solid Tumors
Brief Title: A Study of SGN-CD228A in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed due to portfolio prioritization
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN228-001
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Cutaneous Melanoma; Pleural Mesothelioma; HER2 Negative Breast Neoplasms; Non-small Cell Lung Cancer; Colorectal Cancer; Pancreatic Ductal Adenocarcinoma
Keywords: HER2-negative breast cancer; Seattle Genetics
MeSH Terms: conditions — Melanoma; Mesothelioma, Malignant; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SGN-CD228A (Experimental): SGN-CD228A monotherapy
  Interventions: Drug: SGN-CD228A

INTERVENTIONS:
Drug: SGN-CD228A — SGN-CD228A administered into the vein (IV; intravenously)

SUMMARY:
This trial will study SGN-CD228A to find out whether it is an effective treatment for different kinds of cancer. It will also look at what side effects (unwanted effects) may occur. The study will have two parts. Part 1 of the study will find out how much SGN-CD228A should be given for treatment and how often. Part 2 of the study will use the dose found in Part 1 and look at how safe and effective the treatment is.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety, tolerability, PK, and antitumor activity of SGN-CD228A in select advanced solid tumors. The study will include dose escalation and dose expansion, with multiple disease-specific expansion cohorts.

ELIGIBILITY:
Inclusion Criteria

* Metastatic or unresectable solid malignancy that is histologically or cytologically confirmed to be one of the tumor types listed below. Participants must have relapsed, refractory, or progressive disease (PD) and should have no appropriate standard therapy available. Disease-specific escalation/expansion includes the following tumor types.

  * Metastatic cutaneous melanoma(MCM):

    * Metastatic or advanced cutaneous melanoma, excludes acral or mucosal varieties.
    * Participants must have received at least 1 PD-1-targeted therapy unless contraindicated.
    * Participants with targetable mutations should have received at least 1 therapy targeting that mutation unless contraindicated.
  * Malignant pleural mesothelioma (MPM):

    * Participants must have received cisplatin and pemetrexed unless contraindicated.
  * Advanced HER2-negative breast cancer:

    * Participants must have received 1 or more prior lines of therapy for locally advanced or metastatic disease. Prior therapies must include taxane.
    * Hormone-receptor-positive subjects should have received CDK4/6 inhibitor therapy and have received at least 1 prior hormonally-directed therapy, unless contraindicated.
  * Advanced non-small cell lung cancer (NSCLC):

    * Participants must have locally advanced or metastatic EGFR wild-type NSCLC.
    * Participants must have received platinum-based therapy and at least 1 PD-1- or PD-L1-targeted therapy as a single agent or as part of a combination unless contraindicated.
  * Advanced colorectal cancer:

    * Participants must have received 2 or more prior lines of therapy for locally advanced or metastatic disease, including targeted therapies as appropriate.
  * Advanced pancreatic ductal adenocarcinoma (PDAC):

    * Participants must have unresectable or advanced PDAC.
    * Participants must have received 1 or more prior line of therapy for locally advanced or metastatic disease unless contraindicated.
* Participants should be able to provide adequate tumor tissue for biomarker analysis
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Measurable disease per Response Evaluation Criteria for Solid Tumors version 1.1 (RECIST v1.1)

Exclusion Criteria

* History of another malignancy within 3 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death.
* Pre-existing neuropathy Grade 2 or greater
* Retinal or macular disease requiring treatment or ongoing active monitoring
* Prior receipt of SGN-CD228A or MMAE-containing agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to approximately 3.5 years
  Any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Number of participants with laboratory abnormalities | Up to approximately 3.5 years
Number of participants with dose limiting toxicities | Up to approximately 3.5 years

SECONDARY OUTCOMES:
Best response per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to approximately 3.5 years
Best response per modified RECIST (mRECIST) (participants with pleural mesothelioma only) | Up to approximately 3.5 years
Objective response rate (ORR) | Up to approximately 3.5 years
  A participant is determined to have an OR if they achieve a complete response (CR) or partial response (PR) after initiation of study treatment and at or prior to the end-of-treatment disease assessment.
Progression-free survival (PFS) | Up to approximately 3.5 years
  Defined as the time from the start of study treatment to first documentation of disease progression or death due to any cause, whichever comes first.
Overall survival (OS) | Up to approximately 3.5 years
  Defined as the time from the start of any study treatment to the date of death due to any cause.
Duration of objective response (DOR) | Up to approximately 3.5 years
  Defined as the time from start of the first documentation of objective tumor response (complete response [CR] or partial response [PR]) to the first documentation of confirm tumor progression or death due to any cause, whichever comes first.
Duration of complete response | Up to approximately 3.5 years
  Defined as the time from start of the first documentation of CR to the first documentation of confirmed tumor progression or to death due to any cause, whichever comes first.
Maximum concentration (Cmax) of antibody-conjugated monomethylauristatin E (acMMAE) | Up to approximately 3.5 years
Cmax of free MMAE | Up to approximately 3.5 years
Cmax of total antibody | Up to approximately 3.5 years
Time to maximum concentration (Tmax) of acMMAE | Up to approximately 3.5 years
Tmax of free MMAE | Up to approximately 3.5 years
Tmax of total antibody | Up to approximately 3.5 years
Area under the plasma concentration-time curve from time 0 to the last available [AUC (0-last)] of acMMAE | Up to approximately 3.5 years
AUC(0-last) of free MMAE | Up to approximately 3.5 years
AUC(0-last) of total antibody | Up to approximately 3.5 years
Trough concentration (Ctrough) of acMMAE | Up to approximately 3.5 years
Ctrough of free MMAE | Up to approximately 3.5 years
Ctrough of total antibody | Up to approximately 3.5 years
Incidence of anti-drug antibodies (ADA) | Up to approximately 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Anu Gupta, MD, Study Director — Seagen Inc.
Locations (14):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - University of Chicago Medical Center, Chicago, Illinois
  - Wake Forest Baptist Medical Center / Wake Forest University, Winston-Salem, North Carolina
  - Case Western Reserve University / University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Medical Center (UPMC)/Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
- Institut Gustave Roussy, Villejuif, France
- Istituto Europeo di Oncologia, Milan, Italy
- Hospital Universitario Vall d'Hebron, Barcelona, Spain
- The Royal Marsden Hospital (Surrey), Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mazahreh R, Mason ML, Gosink JJ, Olson DJ, Thurman R, Hale C, Westendorf L, Pires TA, Leiske CI, Carlson M, Nguyen LT, Cochran JH, Okeley NM, Yumul R, Jin S, Stone IJ, Sahetya D, Nesterova A, Allred S, Hensley KM, Hu R, Lawrence R, Lewis TS, Sandall S. SGN-CD228A Is an Investigational CD228-Directed Antibody-Drug Conjugate with Potent Antitumor Activity across a Wide Spectrum of Preclinical Solid Tumor Models. Mol Cancer Ther. 2023 Apr 3;22(4):421-434. doi: 10.1158/1535-7163.MCT-22-0401. PMID 36800443